CLINICAL TRIAL: NCT04352049
Title: Comparing the Dynamics of Changes in Regional Cerebral Oxygen Saturation With Arterial Oxygen Partial Pressure With Two Techniques of Preoxygenation in Healthy Adults
Brief Title: Assessment Through Transcutaneous Brain Oximetry (NIRS) of Two Preoxygenation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, Manuel Ángel Gómez-Ríos, Anesthesiologist, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: JCG-PTO-2012
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia; Functional
Keywords: airway management; general anaesthesia; standard of care; respiration; neurophysiological monitoring.
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3TV group (Active Comparator): Patients were randomly assigned to receive either three minutes tidal volume (3TV) with a fresh gas flow (FGF 100% O2) via facemask of 5 L/min
  Interventions: Procedure: Preoxygenation
- 8DB group (Active Comparator): Or eight vital capacity breaths for 1 minute with FGF of 10 L/min
  Interventions: Procedure: Preoxygenation

INTERVENTIONS:
Procedure: Preoxygenation

SUMMARY:
Preoxygenation techniques is currently considered a standard of care, but how they influence cerebral oxygenation remains largely unknown. In this study, the investigators compare three minutes tidal volume breathing versus eight vital capacity, deep breaths (8DB) technique. Forty-eight patients scheduled for surgery under general anesthesia were included in a randomized study design. The main endpoints were arterial partial pressure of O2 (PaO2) and regional cerebral oxygen saturation (rScO2 ; INVOS TM -5100- C) which were measured at baseline (T1), end of pre-oxygenation (T2) and after desaturation during apnoea to 95% (T3).

DETAILED DESCRIPTION:
Hypoxemia secondary to the inability to secure the airway remains the main cause of anesthesia-related morbidity and mortality. Preoxygenation with 100% oxygen before induction of anesthesia is currently considered a standard of care and practiced routinely for all patients, and especially carefully for high-risk cases. It is an essential component of the rapid sequence induction technique.

Common pre-oxygenation techniques include the 3 min tidal volume breathing (3TV) and the eight vital capacity, deep breaths (8DB). Their efficiency has been extensively assessed by measuring the rate of decline of SaO2 during apnea after induction/paralysis, with 'time to desaturation (to 95% or 90%) being the endpoint of many studies. This is arguably a surrogate endpoint for oxygen stores and Pandit et al. estimated the total amount of oxygen taken up by the body in these techniques using breath-by-breath gas analysis. An even more relevant measure is the impact of preoxygenation on tissue stores of oxygen, but this is difficult to quantify. Especially, given its vulnerability to hypoxemia due to its high energy requirements compared to the low energy reserves, the brain is particularly susceptible.

Cerebral oximetry is a noninvasive monitoring technique that uses near-infrared spectroscopy (NIRS) to measure regional cerebral oxygen saturation (rScO2). Continuous rScO2 monitoring has shown to be useful in detecting mismatch of oxygen supply and demand in the brain and assessing cerebral autoregulation in real-time. This offers a means to measure tissue oxygenation in a relevant organ with pre-oxygenation.

The primary aim of the present study was to test the hypothesis that different pre-oxygenation techniques result in different degrees of cerebral oxygenation as measured by rScO2 with the INVOSTM-5100-C. The investigators wished to compare the 3TV method with the 8DB method, as being the two methods that produced the highest increases in body oxygen stores in previous experiments; the null hypothesis that these would yield similar degrees of brain oxygenation. The investigators also wished to assess whether, regardless of the preoxygenation technique, there were differences between arterial PO2 and rScO2 dynamics with preoxygenation and subsequent apnoea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients scheduled for surgery under general anaesthesia with tracheal intubation
* ASA physical status 1
* aged between 18 and 65 years.

Exclusion Criteria:

* Baseline peripheral oxygen saturation (SpO2) of less than 95%,
* BMI > 30 kg.m-2,
* cardiac, respiratory or brain diseases,
* previous or active smoking,
* predicted difficult airway,
* frontal sinusitis,
* cerebral vascular disorders,
* hemoglobin less than 13g.dL-1,
* low-quality rScO2 signal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-04-15 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2014-10-15 (Actual)

PRIMARY OUTCOMES:
Cerebral regional oxygen saturation (rScO2) | Preoxygenation period, an average of 10 minutes
  rScO2 using an INVOSTM 5100C monitor (Somanetics Corporation, Michigan, USA) and Adult SomaSensor® SAFB-SM sensors (Covidien LLC, MA, USA) placed according to the manufacturers' instructions.

SECONDARY OUTCOMES:
pO2 | Preoxygenation period, an average of 10 minutes
  partial pressure of oxygen through samples for arterial blood gas analyses using the GEM® Premier 3000 monitor (Instrumentation Laboratory. Lexington, MA, USA).
pCO2 | Preoxygenation period, an average of 10 minutes
  partial pressure of CO2 through samples for arterial blood gas analyses using the GEM® Premier 3000 monitor (Instrumentation Laboratory. Lexington, MA, USA).
bispectral index (BIS) | Preoxygenation period, an average of 10 minutes
  by means of a BIS VISTATM monitor (Aspect Medical Systems Inc, Massachusetts, USA)
Cardiac index (CI) | Preoxygenation period, an average of 10 minutes
  using a VigileoTM monitor (Edwards Lifesciences LLC. Irvine, USA
continuous intra-arterial blood pressure | Preoxygenation period, an average of 10 minutes
  . A 20-G cannula was placed in the left radial artery to obtain continuous intra-arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Garzón, MD, Study Director — Complejo Asistencial Salamanca
Locations (2):
- Spain (2):
  - Manuel Gómez-Ríos, A Coruña, Galicia
  - Complexo Hospitalario Universitario de A Coruña, A Coruña

REFERENCES:
- [Background] Joffe AM, Aziz MF, Posner KL, Duggan LV, Mincer SL, Domino KB. Management of Difficult Tracheal Intubation: A Closed Claims Analysis. Anesthesiology. 2019 Oct;131(4):818-829. doi: 10.1097/ALN.0000000000002815. PMID 31584884
- [Background] Baillard C, Boubaya M, Statescu E, Collet M, Solis A, Guezennec J, Levy V, Langeron O. Incidence and risk factors of hypoxaemia after preoxygenation at induction of anaesthesia. Br J Anaesth. 2019 Mar;122(3):388-394. doi: 10.1016/j.bja.2018.11.022. Epub 2018 Dec 29. PMID 30770057
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Pandit JJ. The analysis of variance in anaesthetic research: statistics, biography and history. Anaesthesia. 2010 Dec;65(12):1212-20. doi: 10.1111/j.1365-2044.2010.06542.x. PMID 21182603